CLINICAL TRIAL: NCT04202237
Title: Using the Speckle Doppler to Quantify Perfusion Quality in Kidney and Pancreas Grafts on Vascular Reperfusion
Brief Title: Using the Speckle Doppler to Quantify Blood Flow in Kidney and Pancreas Grafts
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00075
Record Dates: First submitted 2019-12-11; First posted 2019-12-17 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Kidney Transplant Failure and Rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Laser Speckle Contrast Imaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and cell pellets following blood centrifugation will be collected and stored.
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Other: Speckle Doppler imaging — Speckle Doppler Laser imaging
  Other Names: Laser Imaging
Other: Blood sample — Blood sampling
  Other Names: Venepuncture

SUMMARY:
Kidney and Pancreas transplantation is considered the treatment of choice for many people with End Stage Renal Disease and Type 1 diabetes because quality of life and survival is often better after transplantation. However the quality of organs varies as does the quality of perfusion once they are transplanted. The immediate determinant of the survival of any transplanted allograft often depends on the overall quality of perfusion of the organ. The assessment of perfusion is currently visually and empirically done and reported by the surgical team, with low objectivity. The Laser Speckle Doppler technique will be used in both kidney and pancreas transplantation to objectively study the quality of blood flow to the kidney and pancreas after transplantation. This Doppler will provide continuous, non-invasive blood flow monitoring of the microvascular environment of the transplanted organ. The strength of the technique is in evaluating changes in flow over an area of interest or the whole transplanted organ and accurately numerically quantifying the flow. The laser speckle Doppler technique is now well established and has been used in various clinical and research setting as the most convenient means of assessing tissue blood flow. It has however not yet been used in kidney and pancreas transplantation.

DETAILED DESCRIPTION:
BACKGROUND After reperfusion in solid organ transplantation, the quality of organ reperfusion is often assessed visually and reported as good, moderate, reasonable, patchy or poor. In our centre a Renogram is usually performed which uses radioactive tracer which most kidney transplant recipients would have within 24 hours after transplantation to assess the overall perfusion of the allograft. The Speckle Laser Doppler is a powerful clinical tool to obtain full field, high resolution images of microvascular perfusion of an organ It has been used in many medical fields such as dermatology vascular medicine and neurosciences both in a research and in clinical settings. This study seeks to utilise this technique to try to accurately quantify perfusion in the kidney and pancreas after transplantation and to develop a robust numerical quantification system of reporting on organ perfusion.

The Speckle Laser Doppler blood flow imager uses the laser speckle contrast technique to deliver real-time blood flow images with numerical physical data, providing outstanding performance in a wide range of pre-clinical and clinical research applications. This technique has not yet been applied for the assessment of kidney transplant perfusion reporting.

RESEARCH QUESTION/AIM(S)

1. To evaluate the use of the laser blood flow imager in both kidney and pancreas transplantation and obtain real time video images with physical parametric data of the blood flow of transplanted organs at the time of transplantation as a proof of principle study to accurately quantify the blood flow rate either in the whole transplanted organ or a specific area of interest so as to develop a robust numerical quantification system of reporting on the perfusion of the transplanted organ. While this technique has been used in neurosurgery and other clinical settings it has not been evaluated before in a transplant setting.

   .
2. Measure the markers of inflammation (Hypo perfusion) and oxidative stress and attempt correlation with the quality of perfusion obtained.

Objectives

This study aims to utilise this technique to try to accurately quantify perfusion in the kidney and pancreas after transplantation and to develop a robust numerical quantification system of reporting on organ perfusion

Outcome Circulating markers of hypo perfusion and kidney injury will be measured to include: lactate, glutamate, pyruvate, Interleukin 6 as well as glutathione a marker of oxidative stress and assess their correlation with outputs from the two devices.

RATIONALE This study seeks to utilise this technique to try to accurately quantify perfusion in the kidney and pancreas after transplantation and to develop a robust numerical quantification system of reporting on organ perfusion.

The moorFLPI-2 blood flow imager uses the laser speckle contrast technique to deliver real-time blood flow images with numerical physical data, providing outstanding performance in a wide range of pre-clinical and clinical research applications. This technique has not yet been applied for the assessment of kidney transplant perfusion reporting.

STUDY DESIGN and METHODS of DATA COLLECTION AND DATA ANALYIS Speckle Doppler The Speckle Laser Doppler blood flow imager will be used to obtain real-time blood flow images at reperfusion and immediately thereafter this imaging will occur immediately after the surgery when the patient is still under anaesthetic it will take approximately 15 minutes. Initially these images with the flow parametric data will be stored on a laptop which comes with the rental equipment. However once the study is complete, all images and data will be stored on a desktop/drive in the department along with other departmental research data confidentially. The software integrated in the equipment incorporates multiple blood flow parameters and a statistical analytical package for an exhaustive analysis of various parameters. The Speckle Laser Doppler has two low power visible aiming lasers that indicate the approximate centre of the image. The aiming lasers will appear as a single point at a distance of 25 cm. As the distance is increased or decreased from 25 cm, the aiming lasers will appear as two separate points with the centre of the image being located at the midpoint between them. The aiming lasers can be turned on or off by pressing the button on the scan head or from the System Setup window in the PC software.

The moorFLPI-2 measurement software provides two measurement modes that can be used separately or in combination:

* Multi-image measurement mode.
* Single point measurement mode. The multi-image mode setting will be used as it measures flux over regular timed intervals and that is what is required for us to quantify the perfusion as compared to a single point measurement mode which measures the average flux at a single point in time.

Blood samples Concurrently blood samples will be obtained on each patient on Day 0 (day of transplantation), after reperfusion to measure markers of hypo perfusion and kidney injury: lactate, glutamate, pyruvate, Interleukin 6 as well as glutathione a marker of oxidative stress

Clinical Follow up

Patients will be monitored for 3 years following their transplant to look for any transplant related problems which may relate to the quality of the organ as assessed by speckle Doppler.

Sample size and Statistical analysis This is an exploratory study to evaluate the use of Doppler in kidney transplants and as such sample size is mainly dictated by pragmatic considerations and what is available for the duration of hiring the device. Nevertheless sample of 68 is sufficient to provide reasonable precision for the agreement and correlation tests intended for this study in an exploratory level. The analyses will be mainly descriptive. Tests will be exploratory and in the view of generating information for future larger studies.

Research Q1 The software integrated in the equipment incorporates multiple blood flow parameters and a statistical analytical package for an exhaustive analysis of various parameters. The comparison between the 2 methods for measuring blood flow will be assessed for agreement using the appropriate statistical methodology.

The continuous variables for markers of inflammation, circulating markers of hypo perfusion and oxidative stress will also be assessed for any correlation with speckle Doppler perfusion measurements.

Events at the end of 3 years follow up will be compared with the blood flow measurements in categorical analysis.

STUDY SETTING Our unit performs the largest number of kidneys transplants in the UK so has access to a large number of samples for this project.

All members of the team have academic track records and participate in several on-going research projects. Current research projects are investigating cardiovascular disease, kidney perfusion, and MR imaging.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

Kidney Transplant Recipients

* Age between 18 and 75 years
* English Speaking as no funding for translators available
* Able to provide written informed consent
* Receiving a kidney transplant at Manchester University NHS Foundation Trust

Pancreas Transplant Recipients

* Age between 18 and 75 years
* English Speaking as no funding for translators available
* Able to provide written informed consent All individuals will be considered for inclusion in this study regardless of age, disability, gender reassignment, marriage and civil partnership, pregnancy and maternity, race, religion and belief, sex, and sexual orientation except where the study inclusion and exclusion criteria EXPLICITLY state otherwise.

Exclusion Criteria:

Exclusion criteria

* Outside of stated age range. Aged 76+

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study plans to recruit all recipients of, both kidney and pancreas transplants within a 14-week course of the study (Period of Lease of the Speckle Laser Doppler).
  It is expected that approximately n=60 kidney transplants (Living Donor, DBD and DCD and Marginal Kidneys) and n=8 pancreas transplant patients will be recruited in this study period.
  This will provide a range of grafts of varying quality of perfusion for assessment
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the use of the laser blood flow imager in both kidney and pancreas transplantation | 3 months
  Doppler imaging of kidneys and pancreas

SECONDARY OUTCOMES:
Measure the markers of inflammation ng/ml Hypo perfusion and oxidative stress (ng/ml) and attempt correlation with the quality of perfusion obtained | 6-12 months
  Circulating biomarkers of inflammation and oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Titus Augustine, FRCS, Principal Investigator — Manchester university foundation Trust
Locations (1):
- Manchester University NHS Foundationn Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gopal JP, Vaz O, Varley R, Spiers H, Goldsworthy MA, Siddagangaiah V, Lock B, Sharma V, Summers A, Moinuddin Z, van Dellen D, Augustine T. Using Laser Speckle Contrast Imaging to Quantify Perfusion Quality in Kidney and Pancreas Grafts on Vascular Reperfusion: A Proof-of-Principle Study. Transplant Direct. 2023 Apr 19;9(5):e1472. doi: 10.1097/TXD.0000000000001472. eCollection 2023 May. PMID 37090123